CLINICAL TRIAL: NCT05585957
Title: THE VALUE OF INTERLEUKIN 6 AS A DIAGNOSTIC MARKER IN NEONATAL SEPSIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Doha Faisal Hamdallah, Resident of clinical and chemical pathology department, Sohag university hospital, Sohag University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-22-10-08
Record Dates: First submitted 2022-10-16; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: NEONATAL SEPSIS
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: INTERLEUKIN 6 — role of interleukin 6 in the diagnosis of neonatal sepsis in comparison with the routine diagnostic markers of neonatal sepsis

SUMMARY:
Neonatal sepsis is a leading cause of neonatal mortality and continues to be a formidable problem for neonatologists and pediatricians world over. The prevalence of neonatal sepsis varies in different countries; in developed countries it is 1 to 10 cases per 1000 live births and in developing countries the incidence of neonatal septicemia increases to 49 to 170 cases per 1000 live births. The normal fetus is sterile until shortly before birth as the placenta and amniotic sac are highly effective barriers to infections. At birth, the newborn loses the protection afforded to it in the uterus and gets exposed to the microbial world.Neonatal sepsis is broadly divided into two types according to age of onset: Early-onset sepsis (<72 Hrs) and late-onset sepsis (≥72 hrs-28 days). Early-onset sepsis is acquired during fetal life, delivery, or at the nursery.Bacterial organisms causing NS may differ among countries, however, in most developing countries, gram-negative bacteria remain the major source of infection.To date, blood culture is the gold standard test for diagnosing sepsis, but it has some inherent limitations. It takes at least three or five days to be decisive and can be mistakenly negative because antibiotics are initiated empirically before collection and a well-developed microbiology laboratory is required.CRP is one of the most widely studied and applied acute phase proteins clinically, which can be induced by pre-inflammatory factor interleukin-6 (IL-6) to synthesize by liver cells, and it starts to rise in 12-24 hours of inflammatory response and reaches its peak at 48 hours.Interleukin-6 (IL-6) is a pleiotropic cytokine expressed by different cells in response to infections.

ELIGIBILITY:
Inclusion Criteria:

- Neonates admitted to our hospital NICU with fever, poor feeding and irritability whom suspected to have neonatal sepsis.

Exclusion Criteria:

* Normal white blood cell count, patients whom on antibiotic therapy, negative blood culture

Ages: 1 Hour to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
level of interleukin 6 | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guo J, Luo Y, Wu Y, Lai W, Mu X. Clinical Characteristic and Pathogen Spectrum of Neonatal Sepsis in Guangzhou City from June 2011 to June 2017. Med Sci Monit. 2019 Mar 29;25:2296-2304. doi: 10.12659/MSM.912375. PMID 30924465
- [Background] Habib A, Raza S, Ali U, Zubairi AM, Salim E. Diagnostic Accuracy of Serum Procalcitonin (PCT) as an Early Biomarker of Neonatal Sepsis using Blood Culture as Gold Standard. J Coll Physicians Surg Pak. 2021 Apr;31(4):383-387. doi: 10.29271/jcpsp.2021.04.383. PMID 33866721
- [Background] Kan B, Razzaghian HR, Lavoie PM. An Immunological Perspective on Neonatal Sepsis. Trends Mol Med. 2016 Apr;22(4):290-302. doi: 10.1016/j.molmed.2016.02.001. Epub 2016 Mar 15. PMID 26993220
- [Background] Liu C, Fang C, He Q, Xie L. The value of interleukin-6 (IL-6) within 6 hours after birth in the prompt diagnosis of early-onset neonatal sepsis. Transl Pediatr. 2020 Oct;9(5):629-635. doi: 10.21037/tp-20-239. PMID 33209725